CLINICAL TRIAL: NCT01760460
Title: A Multicenter, 24-Week, Double-Blind, Randomized, Placebo-Controlled, Phase III Study With 28-Week Open Labeled Extension Period to Assess the Efficacy and Safety of MK-0859 When Added to Ongoing Statin Therapy With or Without Other Lipid Modifying Medication(s) in Japanese Patients With Dyslipidemia
Brief Title: A Study of the Safety and Efficacy of Anacetrapib (MK-0859) When Added to Ongoing Statin Therapy in Japanese Participants With Dyslipidemia (MK-0859-051 AM1)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0859-051; 132236 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — anacetrapib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anacetrapib (Experimental): Participants will receive 100-mg anacetrapib, orally, once-daily for 24 weeks. Participants will continue on once-daily 100-mg anacetrapib during 28 week open-label extension.
  Interventions: Drug: Anacetrapib
- Placebo (Placebo Comparator): Participants will receive placebo tablet, orally, once daily for 24 weeks. Participants will be switched to once-daily 100-mg anacetrapib during 28 week open-label extension.
  Interventions: Drug: Placebo for anacetrapib

INTERVENTIONS:
Drug: Anacetrapib
  Other Names: MK-0859
  Arms: Anacetrapib
Drug: Placebo for anacetrapib
  Arms: Placebo

SUMMARY:
This study will evaluate the effects of anacetrapib (MK-0859) on low-density lipoprotein-cholesterol (LDL-C) when compared to placebo in Japanese participants with dyslipidemia when added to an existing statin-modifying therapy.

ELIGIBILITY:
Inclusion Criteria:

* If female, cannot be of reproductive potential
* Treatment with an appropriate, stable dose of statin ± other lipid modifying therapy for at least 6 weeks and who is not at LDL-C goal per their category in the Japan Atherosclerosis Society guidelines

Exclusion Criteria:

* Previously participated in a study with a cholesteryl ester transfer protein (CETP) inhibitor
* Homozygous and heterozygous familial hypercholesterolemia
* Severe chronic heart failure
* Uncontrolled cardiac arrhythmias, myocardial infarction (MI), percutaneous coronary intervention (PCI), coronary artery by-pass graft (CABG), unstable angina, or stroke within 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2013-03-14 (Actual); Primary Completion 2015-03-04 (Actual); Study Completion 2015-03-04 (Actual)

PRIMARY OUTCOMES:
Percent Change from Baseline in LDL-C (beta-quantification [BQ] method) | Baseline and Week 24
Percentage of Participants who Experience at Least One Adverse Event (AE) | 64 weeks

SECONDARY OUTCOMES:
Percent Change from Baseline in High-density Lipoprotein-cholesterol (HDL-C) | Baseline and Week 24
Percent Change from Baseline in Non-HDL-C | Baseline and Week 24
Percent Change from Baseline in Apolipoprotein B (Apo-B) | Baseline and Week 24
Percent Change from Baseline in Apolipoprotein A-I (Apo-A-I) | Baseline and Week 24
Percent Change from Baseline in Lipoprotein(a) (Lp[a]) | Baseline and Week 24

REFERENCES:
- [Result] Teramoto T, Daida H, Ikewaki K, Arai H, Maeda Y, Nakagomi M, Shirakawa M, Watanabe Y, Kakikawa T, Numaguchi H, Johnson-Levonas AO, Blaustein RO. Lipid-modifying efficacy and tolerability of anacetrapib added to ongoing statin therapy in Japanese patients with dyslipidemia. Atherosclerosis. 2017 Jun;261:69-77. doi: 10.1016/j.atherosclerosis.2017.03.009. Epub 2017 Mar 10. PMID 28478132